CLINICAL TRIAL: NCT04483804
Title: Application of Radiomics in Correlation Between Ultrasound Characteristics and Pathological Prognostic Factors in Breast Cancer
Brief Title: Application of Radiomics in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHZhejiangU---Breast
Record Dates: First submitted 2020-05-13; First posted 2020-07-23 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Ultrasound; Elastography; Pathology; Radiomics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- disease free survival: Time from randomization to relapse or death due to disease progression
  Interventions: Combination Product: Endocrine therapy
- non-disease free survival: Time of metastasis or death
  Interventions: Combination Product: Endocrine therapy

INTERVENTIONS:
Combination Product: Endocrine therapy — Endocrine therapy

SUMMARY:
Little is known about the correlation between ultrasound characteristics (conventional, elastography and contrast enhanced ultrasound (CEUS) )and pathological prognostic factors in breast cancer. The aim of this study was to explore the correlation between ultrasound characteristics and pathological prognostic factors using radiomics.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of breast cancer

Exclusion Criteria:

Missing pathology Missing follow-up results Missing data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female dominated
Study Population: patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
metastasis | through study completion, an average of 1 year
  lymph node metastasis and/or distant metastasis
death | through study completion, an average of 1 year
  death

CONTACTS AND LOCATIONS:
Overall Officials: pintong Huang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- the Second Affiliated Hospital Zhejiang University School of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data (IPD) can be shared after the main unit publish articles
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: by request
Access Criteria: by request